CLINICAL TRIAL: NCT05987449
Title: A Phase I/II Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of NXT007 in Persons With Severe or Moderate Hemophilia A
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of NXT007 in Persons With Severe or Moderate Hemophilia A
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: WP44714; 2023-503906-35-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1: Cohort 1 - NXT007 Dose Level 1 (Low) (Experimental)
  Interventions: Drug: NXT007
- Part 1: Cohort 2 - NXT007 Dose Level 2 (Experimental)
  Interventions: Drug: NXT007
- Part 1: Cohort 3 - NXT007 Dose Level 3 (Experimental)
  Interventions: Drug: NXT007
- Part 1: Cohort 4 - NXT007 Dose Level 4 (Experimental)
  Interventions: Drug: NXT007
- Part 1: Cohort 5 - NXT007 Dose Level 5 (High) (Experimental)
  Interventions: Drug: NXT007
- Part 2: Cohort A - NXT007 (Experimental)
  Interventions: Drug: NXT007

INTERVENTIONS:
Drug: NXT007 — Participants will receive NXT007 administered subcutaneously (SC), 2 loading doses once every two weeks (Q2W) followed by once every 4 weeks (Q4W) maintenance doses based on the schedule.
  Other Names: Zemocimig; RO7589655; RG6512

SUMMARY:
WP44714 is a Phase I/II, open-label, non-randomized, global, multicenter trial consisting of two parts:

* Part 1 is a multiple-ascending dose (MAD) study in adult and adolescent male participants with severe or moderate hemophilia A with or without factor VIII (FVIII) inhibitors.
* Part 2 is a multiple-dose study in pediatric male participants with severe or moderate hemophilia A with or without FVIII inhibitors.

The overall aim of the study is to investigate the safety, tolerability, pharmacokinetics, pharmacodynamics, immunogenicity, and efficacy of NXT007.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe (Factor VIII [FVIII] coagulant activity <1 IU/dL) or moderate (FVIII coagulant activity ≥1 IU/dL and ≤5 IU/dL) congenital hemophilia A with or without inhibitors against FVIII
* Participants with FVIII inhibitors: participants using recombinant activated factor VII (rFVIIa) or willing to switch to rFVIIa as primary bypassing agent for the treatment of breakthrough bleeds, trauma, or procedures
* Historic local FVIII inhibitor test results being available during screening to confirm any previous inhibitor history and current status
* Participants who previously successfully completed immune tolerance induction (ITI) must have done so at least 5 years before screening and must have no evidence of inhibitor recurrence (permanent or temporary) since. FVIII tolerance defined as <0.6 Bethesda unit (BU)/mL (<1.0 BU/mL only for laboratories with an historical sensitivity cutoff for inhibitor detection of 1.0 BU/mL) and in vivo recovery >66%
* Documentation of number and type of bleeding episodes in the last 24 weeks prior to enrollment
* Adequate hematologic function, defined as platelet count ≥100,000 cells/μL and hemoglobin ≥11 g/dL at the time of screening
* Adequate hepatic function defined as total bilirubin ≤1.5× age-adapted upper limit of normal (ULN) (excluding Gilbert syndrome) and both aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3× age-adapted ULN at the time of screening, and no clinical signs or known laboratory/radiographic evidence consistent with cirrhosis. For patients with Gilbert syndrome, bilirubin should be <4 mg/dL or 68.4 umol/L at the time of screening.
* For Part 1 only: Adequate renal function, defined as serum creatinine ≤2.5× age-adapted ULN and calculated creatinine clearance ≥30 mL/min by Cockroft-Gault formula
* For Part 2 only: Adequate renal function, defined as serum creatinine ≤1.5× age-adapted ULN. When the serum creatinine is ≥1.5× ULN, creatinine clearance by Bedside Schwartz formula must be >70 mL/min/1.73m^2.
* Willingness and ability to comply with schedules visits, treatment plans, laboratory tests, and other study procedures

Exclusion Criteria:

* Inherited or acquired bleeding disorders other than congenital hemophilia A
* Ongoing or planned ITI therapy
* Previous or current treatment for thromboembolic disease (with the exception of previous catheter-associated thrombosis for which anti-thrombotic treatment is not currently ongoing) or signs of thromboembolic disease
* At high risk for thrombotic microangiopathy (TMA), including past personal or family history of TMA, in the investigator's judgment
* For Part 1 only: Personal history of ischemic heart disease, cerebrovascular disease, or diabetes mellitus
* For Part 1 only: Strong family history of ischemic heart disease or cerebrovascular disease (i.e., first degree relatives such as parents, full siblings, or children): male relatives diagnosed under the age of 55 years and females under the age of 65 years
* For Part 1 only: Previous or concomitant malignancies or leukemia
* Other conditions (e.g., autoimmune conditions such as Systemic Lupus erythematosus and other systemic inflammatory disorders) that may currently increase the risk of bleeding or thrombosis
* History of clinically significant allergies
* Receipt of any of the following:

  i) An investigational drug to treat or reduce the risk of hemophilic bleeds within 5 half-lives of last drug administration or normalization of targeted parameters (e.g., anti-thrombin), whichever is longer; ii) A non-hemophilia-related investigational drug within last 30 days or 5 half-lives, whichever is shorter; iii) Any other investigational drug currently being administered or planned to be administered; iv) Prior gene therapy or gene therapy planned to be administered; v) Use of systemic immunomodulators (e.g., interferon or rituximab) at enrollment or planned use during the study, with the exception of anti-retroviral therapy to treat HIV.
* Protein C activity, protein S free antigen, or anti-thrombin III activity levels below the lower limit of the reference range at screening
* Known HIV infection with CD4 counts <200 cells/μL
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy and to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to excipient content
* History or presence of an abnormal ECG that is deemed clinically significant, (e.g., complete left bundle branch block, second- or third -degree atrioventricular heart block), including atrial fibrillation or evidence of prior myocardial infarction
* QT interval corrected through use of Fridericia's formula (QTcF) >450 ms demonstrated by at least two ECGs >30 minutes apart
* History of ventricular dysrhythmias or risk factors for ventricular dysrhythmias such as structural heart disease (e.g., severe left ventricular systolic dysfunction, left ventricular hypertrophy), coronary heart disease (symptomatic or with ischemia demonstrated by diagnostic testing), clinically significant electrolyte abnormalities (e.g., hypokalemia, hypomagnesemia, hypocalcemia), or family history of sudden unexplained death or long QT syndrome
* Current treatment with medications that are well known to prolong the QT interval

Ages: 2 Years to 59 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2030-06-16 (Estimated); Study Completion 2030-06-16 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Adverse Events, with Severity Determined According to National Cancer Institute Common Terminology Criteria for Adverse Events Grading Scale | From Baseline until study completion or discontinuation (up to 7.5 years)
Number of Participants with at Least One Clinical Laboratory Test Abnormality for Hematology Parameters | From Baseline until study completion or discontinuation (up to 7.5 years)
Number of Participants with at Least One Clinical Laboratory Test Abnormality for Blood Chemistry Parameters | From Baseline until study completion or discontinuation (up to 7.5 years)
Number of Participants with at Least One Vital Sign Abnormality | From Baseline until study completion or discontinuation (up to 7.5 years)
  The vital signs that will be assessed are body temperature, pulse rate, respiratory rate, and systolic and diastolic blood pressure.
Number of Participants with at Least One Abnormality on Electrocardiogram (ECG) Recordings | From Baseline until study completion or discontinuation (up to 7.5 years)
  The ECG parameters that will be assessed are heart rate, PR interval, QRS interval, QT interval, and QTcF inteval.

SECONDARY OUTCOMES:
Plasma Concentration of NXT007 at Specified Timepoints | At prespecified timepoints from Week 1 to Week 23, every 28 days from Week 25 until Week 49, and every 12 weeks thereafter until study completion or discontinuation (up to 7.5 years)
Maximum Observed Plasma Concentration (Cmax) of NXT007 After the First Dose | At prespecified timepoints from Day 1 to Day 15
Time to Maximum Observed Plasma Concentration (tmax) of NXT007 After the First Dose | At prespecified timepoints from Day 1 to Day 15
Area Under the Plasma Concentration-Time Curve (AUC) of NXT007 After the First Dose | At prespecified timepoints from Day 1 to Day 15
Number of Participants Testing Positive for Anti-Drug Antibodies Against NXT007 at Baseline and During Treatment with Study Drug | Baseline (predose on Day 1) and from first dose of study drug until study completion or discontinuation (up to 7.5 years)
Number of Participants Testing Positive for Anti-Factor VIII Inhibitors at Baseline and During Treatment with Study Drug | Baseline (predose on Day 1) and from first dose of study drug until study completion or discontinuation (up to 7.5 years)
Model-Based Annualized Bleeding Rate for Treated Bleeds | From first dose of study drug until study completion or discontinuation (up to 7.5 years)
Mean Calculated Annualized Bleeding Rate for Treated Bleeds | From first dose of study drug until study completion or discontinuation (up to 7.5 years)
Median Calculated Annualized Bleeding Rate for Treated Bleeds | From first dose of study drug until study completion or discontinuation (up to 7.5 years)
Model-Based Annualized Bleeding Rate for All Bleeds | From first dose of study drug until study completion or discontinuation (up to 7.5 years)
Mean Calculated Annualized Bleeding Rate for All Bleeds | From first dose of study drug until study completion or discontinuation (up to 7.5 years)
Median Calculated Annualized Bleeding Rate for All Bleeds | From first dose of study drug until study completion or discontinuation (up to 7.5 years)
Model-Based Annualized Bleeding Rate for Treated Spontaneous Bleeds | From first dose of study drug until study completion or discontinuation (up to 7.5 years)
Mean Calculated Annualized Bleeding Rate for Treated Spontaneous Bleeds | From first dose of study drug until study completion or discontinuation (up to 7.5 years)
Median Calculated Annualized Bleeding Rate for Treated Spontaneous Bleeds | From first dose of study drug until study completion or discontinuation (up to 7.5 years)
Model-Based Annualized Bleeding Rate for Treated Joint Bleeds | From first dose of study drug until study completion or discontinuation (up to 7.5 years)
Mean Calculated Annualized Bleeding Rate for Treated Joint Bleeds | From first dose of study drug until study completion or discontinuation (up to 7.5 years)
Median Calculated Annualized Bleeding Rate for Treated Joint Bleeds | From first dose of study drug until study completion or discontinuation (up to 7.5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- United States (4):
  - UC Davis Cancer Center, Sacramento, California
  - Georgetown Uni Medical Center, Washington D.C., District of Columbia
  - Indiana Hemophilia & Thrombosis center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clnics Dept of Pediatrics, Iowa City, Iowa
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
- Istituto Clinico Humanitas, Rozzano (MI), Lombardy, Italy
- Auckland Cancer Trial Centre, Auckland, New Zealand
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Gda?sk
  - Instytut Hematologii i Transfuzjologii, Warsaw
- Spain (3):
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona
  - Hospital Universitario la Paz, Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga

IPD SHARING:
Plan to Share IPD: No
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing